CLINICAL TRIAL: NCT02281643
Title: Comparison of Early and Late Administration of Doxycycline in Their Efficacy Against Mansonella Perstans and in Development of Immunity Against Mycobacterial Infections
Brief Title: Concomitant Infections of Mansonella Perstans in Tuberculosis and Buruli Ulcer Disease Patients From Ghana
Acronym: Map2Co
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kwame Nkrumah University of Science and Technology (Other)
Collaborators: University of Bonn (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr Richard Phillips, Dr, Kwame Nkrumah University of Science and Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GZ:JA 1479/5-1
Record Dates: First submitted 2014-10-26; First posted 2014-11-03 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Mansonella Perstans Infection; Buruli Ulcer; Tuberculosis; Co-infection
Keywords: Coinfection; Buruli ulcer; Tuberculosis; Mansonella perstans
MeSH Terms: conditions — Mansonelliasis; Buruli Ulcer; Tuberculosis; Coinfection; Dipetalonema Infections | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early doxycycline administered (Experimental): Early doxycycline administered - volunteers will be treated immediately with 200mg daily doxycycline for 6 weeks
  Interventions: Drug: Doxycycline
- Delayed doxycycline administered (Active Comparator): Delayed doxycycline administered-volunteers will be treated six months after the early group has received treatment with 200mg daily doxycycline for 6 weeks
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — 200mg oral doxycycline will be administered immediately (early) in the experimental arm or delayed in the comparator arm
  Other Names: Vibramycim; Oracea

SUMMARY:
This study will determine the influence of doxycycline treatment against Wolbachia/M. perstans on immunity against concomitant mycobacterial infections in healthy M. perstans infected individuals. In this regard, the investigators will perform a community-based randomized controlled trial (Phase 2a) in Asante Akim North District. A cohort of 200 participants who are contacts of patients with Tuberculosis or Buruli ulcer, of both sexes with no clinical condition requiring long-term medication but connected with Mansonella perstans will be investigated for the effect of doxycycline on microfilaria, the immune response and development of mycobacterial disease.

DETAILED DESCRIPTION:
The purpose of this study is to describe the immune response to Mansonella perstans with or without doxycycline treatment. And to suggest the use of doxycycline for the treatment of Mansonella perstans infected individuals. Two hundred Mansonella perstans infected individuals who are contacts of patients with Buruli ulcer or Tuberculosis will be recruited and placed in two groups. Hundred patients in each group ('early', or 'delayed' doxycycline-treatment group) with weight 40kg and above. Individuals will be recruited from communities in the Asante Akim North District.

Half of the M. perstans infected individuals (randomly selected) will be treated immediately with 200mg daily doxycycline for six weeks. All recruited individuals will be asked to donate 20ml; 10 ml heparinized blood, 5ml Ethylenediaminetetraacetic acid blood and 5ml blood for serum analysis at baseline (day 0), after 4 months (day 112), after 12 months (day 336) and after 24 months (day 672). Six months after doxycycline treatment for M. perstans infected individuals the other 100 patients who are not treated at time point 0 (delayed' treatment group) will be treated as described for the 'early' treatment group. After four months (day 112) individuals from both treatment groups will be asked to donate blood for quantitative Polymerase Chain Reaction to confirm Wolbachia depletion and immunological analyses.

For 'early', and 'delayed', doxycycline-treatment group immunological assays will be performed at days 0, 112, 336 and 672 after treatment initiation for all recruited individuals.

Hypothesis:

Presence of filarial nematodes Mansonella perstans will polarize the host immunity towards humoral and T helper type 2-mediated immunity and treatment with doxycycline will result in killing of Wolbachia endosymbionts, depletion of Mansonella perstans and development of a T helper type 1 immunity and reduced risk of developing Tuberculosis and Buruli ulcer

Sample size justification Since the study is a pilot study to gain first experience regarding the primary and secondary endpoints under the intended treatment regimens, the sample size cannot be justified by a statistical argumentation. A sample size of 100 participants (80 participants plus 20% drop-out rate) per treatment arm was chosen in agreement with the study statistician.

Statistical methods The detailed plan for data analysis will be written and discussed with the DMEC before final de-blinding of the data.

Data safety Electronic data will be secured and password limited to persons named in this Study Protocol. Analyses of the data will be performed on copies of the original data files ensuring raw data accessibility at all times. Regular backups to an external hard drive will be carried out ensuring protection against data loss.

Data Monitoring and Ethics Committee (DMEC) Independent monitoring of the clinical trial will be carried out by the DMEC consisting of representatives from key stakeholders in existing filarial control programmes with the necessary expertise covering the range of project activities and skills to provide support and advice on the study progress.

Additionally the External Scientific Advisory Committee (ESAC) will monitor the study ensuring compliance with all directives. DMEC and ESAC members are listed

Informed Consent Form (ICF) Regulatory requirement necessitates obtaining and documenting informed consent, Good Clinical Practice and ethical principles along the Declaration of Helsinki (first adopted 1964, amended five times, most recently in 2000). All consent forms will accompany the study protocol and submitted for approval by the relevant ethic committees.

Patient insurance Professional indemnity liability insurance of the individual volunteers will be obtained to take care of any form of injuries that may arise in the process of drug administration.

ELIGIBILITY:
Inclusion Criteria:

M. perstans mg-positive status Good general health without any clinical condition requiring long-term medication.

Normal renal and hepatic laboratory profiles

Exclusion Criteria:

Known intolerance to the doxycycline Body weight <40 kg Pregnancy or breastfeeding History of severe allergic reaction or anaphylaxis Alcohol or drug abuse

Ages: 9 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Microfilarial assessment | Change from baseline microfilarial load at 12 months
  Assessment of the microfilarial load

SECONDARY OUTCOMES:
Demonstrate development of a T helper type 1 immunity through Immunological profile of cellular immune responses | Change from baseline T helper type 1 cytokine levels at 24 weeks
  Measurement of the T helper type 1 cytokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Richard Phillips O Phillips, MBChB, PhD, Principal Investigator — Kwame Nkrumah University of Science and Technology; Ellis Owusu Dabo, MBChB, PhD, Study Director — Kumasi Centre for Collaborative Research; Alexander Y Debrah, PhD, Study Chair — Kwame Nkrumah University of Science and Technology
Locations (1):
- Agogo Presbyterian Hospital, Agogo, Asante Akim North District, Ghana

REFERENCES:
- [Derived] Debrah LB, Nausch N, Opoku VS, Owusu W, Mubarik Y, Berko DA, Wanji S, Layland LE, Hoerauf A, Jacobsen M, Debrah AY, Phillips RO. Epidemiology of Mansonella perstans in the middle belt of Ghana. Parasit Vectors. 2017 Jan 7;10(1):15. doi: 10.1186/s13071-016-1960-0. PMID 28061905